CLINICAL TRIAL: NCT02497612
Title: A Randomized, Double-blind, Phase IIb Study to Investigate the Efficacy, Safety, Tolerability and Pharmacokinetics of a Single Dose Regimen of Ferroquine (FQ) With Artefenomel (OZ439) in Adults and Children With Uncomplicated Plasmodium Falciparum Malaria
Brief Title: To Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of a Single Dose Regimen of Ferroquine and Artefenomel in Adults and Children With Uncomplicated Plasmodium Falciparum Malaria
Acronym: FALCI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: All treatment arms met the futility criteria for efficacy during the pre-planned interim analysis, therefore the study was stopped.
Sponsor: Sanofi (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRI12805; U1111-1155-7960 (Other: UTN)
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Plasmodium Falciparum Infection
MeSH Terms: interventions — ferroquine; artefenomel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) (Experimental): On Day 0, based on the body weight (BW), participants received orally a single dose of ferroquine (FQ) capsules or oral suspension (along with matching placebo, as applicable to maintain blinding) and a single dose of artefenomel (OZ439) (maximum dose up to 800 milligrams [mg]) oral suspension as follows: BW greater than or equal to (>=) 35 kilograms (kg): FQ 400 mg + OZ439 800 mg; BW >=24 kg to less than (<) 35 kg: FQ 300 mg + OZ439 600 mg; BW >=15 kg to <24 kg: FQ 200 mg + OZ439 400 mg; BW >=10 kg to <15 kg: FQ 150 mg + OZ439 300 mg; BW >=7 kg to <10 kg: FQ 100 mg + OZ439 200 mg; >=5 kg to <7kg: FQ 75 mg + OZ439 150 mg.
  Interventions: Drug: Ferroquine SSR97193; Drug: Artefenomel; Other: Placebo
- Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) (Experimental): On Day 0, based on the BW, participants received orally a single dose of FQ capsules or oral suspension (along with matching placebo, as applicable to maintain blinding) and a single dose of OZ439 (maximum dose up to 800 mg) oral suspension as follows: BW >= 35 kg: FQ 600 mg + OZ439 800 mg; BW >=24 kg to <35 kg: FQ 450 mg + OZ439 600 mg; BW >=15 kg to <24 kg: FQ 300 mg + OZ439 400 mg; BW >=10 kg to <15 kg: FQ 225 mg + OZ439 300 mg; BW >=7 kg to <10 kg: FQ 150 mg + OZ439 200 mg; >=5 kg to <7kg: FQ 115 mg + OZ439 150 mg.
  Interventions: Drug: Ferroquine SSR97193; Drug: Artefenomel; Other: Placebo
- Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) (Experimental): On Day 0, based on the BW, participants received orally a single dose of FQ capsules or oral suspension (along with matching placebo, as applicable to maintain blinding) and a single dose of OZ439 (maximum dose up to 800 mg) oral suspension as follows: BW >= 35 kg: FQ 900 mg + OZ439 800 mg; BW >=24 kg to <35 kg: FQ 675 mg + OZ439 600 mg; BW >=15 kg to <24 kg: FQ 450 mg + OZ439 400 mg; BW >=10 kg to <15 kg: FQ 335 mg + OZ439 300 mg; BW >=7 kg to <10 kg: FQ 225 mg + OZ439 200 mg; >=5 kg to <7kg: FQ 170 mg + OZ439 150 mg.
  Interventions: Drug: Ferroquine SSR97193; Drug: Artefenomel; Other: Placebo
- Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg) (Experimental): On Day 0, based on the BW, participants received orally a single dose of FQ capsules or oral suspension (along with matching placebo, as applicable to maintain blinding) and a single dose of OZ439 (maximum dose up to 800 mg) oral suspension as follows: BW >= 35 kg: FQ 1200 mg + OZ439 800 mg; BW >=24 kg to <35 kg: FQ 900 mg + OZ439 600 mg; BW >=15 kg to <24 kg: FQ 600 mg + OZ439 400 mg; BW >=10 kg to <15 kg: FQ 450 mg + OZ439 300 mg; BW >=7 kg to <10 kg: FQ 300 mg + OZ439 200 mg; >=5 kg to <7kg: FQ 225 mg + OZ439 150 mg.
  Interventions: Drug: Ferroquine SSR97193; Drug: Artefenomel; Other: Placebo

INTERVENTIONS:
Drug: Ferroquine SSR97193 — Pharmaceutical form:Capsules Route of administration: oral
Drug: Artefenomel — Pharmaceutical form:Granules for suspension Route of administration: oral
Other: Placebo — Capsules. Placebo capsules were used to keep the same number of capsules in each weight band while keeping the ferroquine dose blinded. No participant received placebo only.

SUMMARY:
Primary Objective:

To determine whether a single dose combination of OZ439 (Artefenomel)/FQ (Ferroquine) was an efficacious treatment for uncomplicated Plasmodium falciparum malaria in adults and children.

Secondary Objectives:

* To evaluate the efficacy of OZ439/FQ:

  * To determine the incidence of recrudescence and re-infection.
  * To determine the time to relief of fever and parasite clearance.
* To evaluate the safety and tolerability of OZ439/FQ in adults and children.
* To characterize the pharmacokinetics of OZ439 in plasma, FQ and its active metabolite SSR97213 in blood.
* To determine the blood/plasma ratio for FQ and SSR97213 in some participants at limited time points in selected sites.

DETAILED DESCRIPTION:
Total duration was 63 days for each participant.

ELIGIBILITY:
Inclusion criteria:

Male or female participant aged greater than (>) 6 months old and <70 years old:

* Cohort 1 = 14 years < age <70 years and body weight greater than or equal to (>=) 35 kilogram (kg).
* Cohort 2 = 5 years < age less than or equal to (<=) 14 years.
* Cohort 3 = 2 years < age <=5 years.
* Cohort 4 = 6 months < age <=2 years.

Body weight >=5 kg and <=90 kg.

Presence of mono-infection by Plasmodium falciparum with:

* Fever, as defined by axillary temperature >=37.5 degrees Celsius (°C) or oral/rectal/tympanic temperature >=38°C, or history of fever in the previous 24 hours (history of fever must be documented) and,
* Microscopically (blood smear) confirmed parasite infection, ranging from 1000 to 100 000 asexual parasites/microliter of blood.

Informed consent form signed by the participant or by the legally acceptable representative of the minor participant.

Exclusion criteria:

Presence of severe malaria.

Anti-malarial treatment:

* With piperaquine-based compound, mefloquine, naphthoquine or sulphadoxine/pyrimethamine (SP) within the previous 6 weeks (after their inhibition of new infections had fallen below 50%).
* With amodiaquine or chloroquine within the previous 4 weeks.
* With quinine, halofantrine, lumefantrine-based compounds and any other anti-malarial treatment or antibiotics with antimalarial activity (including cotrimoxazole, tetracyclines, quinolones and fluoroquinolones, and azithromycin) within the past 14 days.
* With any herbal products or traditional medicines, within the past 7 days.

Known history or evidence of clinically significant disorders.

Previous treatment within 5 times the half-life or within the last 14 days, whichever the longest which are: P-glycoprotein substrates, Cytochrome P450 (CYP) 2D6 main substrates and/or strong CYP2C or CYP3A inhibitors and/or moderate inhibitors but inhibiting both CYP2C and CYP3A and/or CYP inducers.

Mixed plasmodium infection.

Severe vomiting.

Severe malnutrition.

Laboratory parameters with clinically significant abnormalities and/or reaching critical values. For Liver Function Test. Aspartate aminotransferase (>2 [upper limit of normal] ULN), or alanine aminotransferase (>2 ULN) or total bilirubin >1.5 ULN.

Presence of Hepatitis A Immunoglobulin M, Hepatitis B surface antigen or Hepatitis C antibody.

Had received an investigational drug within the past 4 weeks.

Previous participation in any malaria vaccine study or received malaria vaccine in any other circumstance.

Measles and yellow fever vaccine injection within the last 15 days and or planned for the 28 days after randomization.

Female participant of child bearing potential not willing to use an effective contraceptive(s) method(s) for the duration of the study.

Positive serum or urine beta-human chorionic gonadotropin pregnancy test at study screening for female participants of childbearing potential.

Breastfeeding women.

Male participant having a partner of child bearing potential not willing to use an effective method of birth control during the study treatment period.

Splenectomized participants or presence of surgical scar on left hypochondrium. Participant unable to drink.

Known history of hypersensitivity, allergic or anaphylactoid reactions to ferroquine or other amino-quinolines or to OZ439 or OZ277 or to any of the excipients.

Family history of sudden death or of congenital prolongation of the Corrected QT (QTc) interval or known congenital prolongation of the QTc interval or any clinical condition known to prolong the QTc interval e.g., participants with a history of symptomatic cardiac arrhythmias or with clinically relevant bradycardia.

QTc using Fridericia's formula >450 millisecond at screening or pre-dose.

Hypokalemia (<3.5 millimoles per liter [mmol/L]), hypocalcemia (<2.0 mmol/L) or hypomagnesemia (<0.5 mmol/L) at screening or pre-dose.

Any treatment known to induce a lengthening of QT interval.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 6 Months to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2015-07-25 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (12):
- Investigational Site Number 204001, Cotonou, Benin
- Burkina Faso (3):
  - Investigational Site Number 854002, Comoé
  - Investigational Site Number 854003, Niangoloko
  - Investigational Site Number 854001, Ouagadougou
- Gabon (2):
  - Investigational Site Number 266002, Lambaréné
  - Investigational Site Number 266001, Libreville
- Kenya (2):
  - Investigational Site Number 404003, Kisumu
  - Investigational Site Number 404002, Siaya
- Investigational Site Number 508001, Chokwé, Mozambique
- Investigational Site Number 800002, Tororo, Uganda
- Vietnam (2):
  - Investigational Site Number 704003, Bình Phước
  - Investigational Site Number 704004, Pleiku

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Adoke Y, Zoleko-Manego R, Ouoba S, Tiono AB, Kaguthi G, Bonzela JE, Duong TT, Nahum A, Bouyou-Akotet M, Ogutu B, Ouedraogo A, Macintyre F, Jessel A, Laurijssens B, Cherkaoui-Rbati MH, Cantalloube C, Marrast AC, Bejuit R, White D, Wells TNC, Wartha F, Leroy D, Kibuuka A, Mombo-Ngoma G, Ouattara D, Mugenya I, Phuc BQ, Bohissou F, Mawili-Mboumba DP, Olewe F, Soulama I, Tinto H; FALCI Study Group. A randomized, double-blind, phase 2b study to investigate the efficacy, safety, tolerability and pharmacokinetics of a single-dose regimen of ferroquine with artefenomel in adults and children with uncomplicated Plasmodium falciparum malaria. Malar J. 2021 May 19;20(1):222. doi: 10.1186/s12936-021-03749-4. PMID 34011358

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study conducted at 12 active sites in 7 countries. Total of 806 participants were screened between 25 July 2015 and 22 July 2019, of which 377 were randomized to 1 of 4 treatment arms (via Integrated Web Recognition System using permuted block randomization schedules). 429 participants failed screening mainly due to meeting exclusion criteria.
Pre-assignment Details: In each arm, participants were divided in 4 cohorts (C):C1 (greater than [>] 14 years (yrs) to less than [<] 70 yrs); C2 (>5 yrs to less than or equal to [<=] 14 yrs );C3 (>2 yrs to <=5 yrs); C4 (>6 months to <=2 yrs). Day 0 (drug administration day, per protocol) was Day 1 for safety reporting as per Clinical Data Interchange Standards Consortium.
Groups:
- Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg): On Day 0, based on the body weight (BW), participants received orally a single dose of ferroquine (FQ) capsules or oral suspension (along with matching placebo, as applicable to maintain blinding) and a single dose of artefenomel (OZ439) (maximum dose up to 800 milligrams [mg]) oral suspension as follows: BW greater than or equal to (>=) 35 kilograms (kg): FQ 400 mg + OZ439 800 mg; BW >=24 kg to <35 kg: FQ 300 mg + OZ439 600 mg; BW >=15 kg to <24 kg: FQ 200 mg + OZ439 400 mg; BW >=10 kg to <15 kg: FQ 150 mg + OZ439 300 mg; BW >=7 kg to <10 kg: FQ 100 mg + OZ439 200 mg; >=5 kg to <7kg: FQ 75 mg + OZ439 150 mg.
Period: Overall Study
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Started | 93 | 94 | 97 | 93
Treated | 92 | 94 | 96 | 91
Cohort 1: >14 Years to <70 Years | 14 | 15 | 18 | 16
Cohort 2: >5 Years to <=14 Years | 6 | 5 | 6 | 5
Cohort 3: >2 Years to <=5 Years | 66 | 66 | 67 | 65
Cohort 4: >6 Months to <=2 Years | 7 | 8 | 6 | 7
Completed | 27 | 37 | 48 | 46
Not Completed | 66 | 57 | 49 | 47
Not completed — Met >=1 anti-malarial treatment criteria | 57 | 51 | 39 | 41
Not completed — Participant's request | 2 | 3 | 4 | 1
Not completed — Investigator's judgement | 1 | 0 | 0 | 2
Not completed — Adverse Event | 3 | 1 | 4 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1
Not completed — Other unspecified | 1 | 1 | 2 | 0
Not completed — Not eligible | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg): On Day 0, based on the BW, participants received orally a single dose of FQ capsules or oral suspension (along with matching placebo, as applicable to maintain blinding) and a single dose of OZ439 (maximum dose up to 800 mg oral suspension as follows: BW >= 35 kg: FQ 400 mg + OZ439 800 mg; BW >=24 kg to <35 kg: FQ 300 mg + OZ439 600 mg; BW >=15 kg to <24 kg: FQ 200 mg + OZ439 400 mg; BW >=10 kg to <15 kg: FQ 150 mg + OZ439 300 mg; BW >=7 kg to <10 kg: FQ 100 mg + OZ439 200 mg; >=5 kg to <7kg: FQ 75 mg + OZ439 150 mg.
- Total: Total of all reporting groups
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg) | Total
Number analyzed (Participants) | 93 | 94 | 97 | 93 | 377
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.34 (9.94) | 6.97 (8.97) | 7.61 (9.60) | 7.68 (10.44) | 7.40 (9.71)
Age, Customized [Count of Participants; unit: Participants]
  >6 months to <=2 years | 7 | 8 | 6 | 7 | 28
  >2 to <=5 years | 66 | 66 | 67 | 65 | 264
  >5 to <=14 years | 6 | 5 | 6 | 5 | 22
  >14 to <18 years | 6 | 5 | 7 | 4 | 22
  >=18 years | 8 | 10 | 11 | 12 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 46 | 43 | 56 | 182
  Male | 56 | 48 | 54 | 37 | 195
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 5 | 6 | 6 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 89 | 89 | 91 | 87 | 356
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Polymerase Chain Reaction (PCR)-Adjusted Adequate Clinical and Parasitological Response (ACPR) at Day 28: African <=5 Years Per Protocol Population at Day 28 (PP28)
Description: ACPR: negative parasitemia at Day 28, irrespective of axillary temperature(AT), in participants not meeting any criteria of early therapy failure (ETF):Danger signs (DS)/severe malaria (SM) at Day 1, 2 or 3 in presence of parasitemia; or Day 2 parasite count >Day 0 irrespective of AT; or parasitemia at Day 3 with AT >=37.5 degree Celsius (°C); or parasite count on Day 3>=25 percent (%) on Day 0, or late clinical failure(LCF):DS/ SM in presence of parasitemia between Day 4 and 28; or presence of parasitemia and AT>=37.5°C between Day 4 and 28, or late parasitological failure (LPF):presence of parasitemia between Day 7 and 28 and AT<37.5°C or having rescue therapy for malaria. PCR-adjusted ACPR applied to recrudescence (appearance of asexual parasites after clearance of initial infection with genotype identical to that present at Baseline), excluding participants with re-infection. In data table, "overall number of participants analyzed"=participants evaluable for this outcome measure.
Time Frame: Day 28
Population: African <=5 years PP28: participants with parasitologically confirmed Plasmodium falciparum malaria at screening/baseline, received the single administration of OZ439/FQ, without major protocol violations impacting efficacy, evaluable for crude ACPR at Day 28, excluding those who received rescue treatment due to vomiting during drug administration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 51 | 60 | 57 | 60
percentage of participants | 78.4 [64.7 to 88.7] | 85.0 [73.4 to 92.9] | 89.5 [78.5 to 96.0] | 91.7 [81.6 to 97.2]

2. Secondary Outcome: Percentage of Participants With Polymerase Chain Reaction-adjusted Adequate Clinical and Parasitological Response at Day 28: African >5 Years Per Protocol Population at Day 28 (A5PP28)
Description: ACPR: negative parasitemia at Day 28, irrespective of AT, in participants not meeting any criteria of ETF: DS or SM at Day 1, 2 or 3 in presence of parasitemia; or Day 2 parasite count > Day 0 irrespective of AT; or parasitemia at Day 3 with AT >=37.5°C; or parasite count on Day 3 >=25% on Day 0, or LCF: DS/ SM in presence of parasitemia between Day 4 and 28; or presence of parasitemia and AT >=37.5°C between Day 4 and 28, or LPF: presence of parasitemia between Day 7 and 28 and AT <37.5°C or having rescue therapy for malaria. PCR-adjusted ACPR was applied to recrudescence (appearance of asexual parasites after clearance of initial infection with a genotype identical to that of parasites present at Baseline), excluding participants with re-infection. Here, in the data table, "overall number of participants analyzed"=participants evaluable for this outcome measure.
Time Frame: Day 28
Population: African >5 years PP28: participants with parasitologically confirmed Plasmodium falciparum malaria at screening/baseline, received the single administration of OZ439/FQ, without major protocol violations impacting efficacy, evaluable for crude ACPR at Day 28, excluding those who received rescue treatment due to vomiting during drug administration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 11 | 10 | 12 | 10
percentage of participants | 72.7 [39.0 to 94.0] | 100 [69.2 to 100] | 100 [73.5 to 100] | 90.0 [55.5 to 99.7]

3. Secondary Outcome: Percentage of Participants With Polymerase Chain Reaction-adjusted Adequate Clinical and Parasitological Response at Day 28: Asian PP Population at Day 28 (APP28)
Description: as for outcome 2
Time Frame: Day 28
Population: Asian PP28 population: participants with parasitologically confirmed Plasmodium falciparum malaria at screening/baseline, received the single administration of OZ439/FQ, without major protocol violations impacting efficacy, evaluable for crude ACPR at Day 28, excluding those who received rescue treatment due to vomiting during drug administration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 4 | 4 | 5 | 5
percentage of participants | 25.0 [0.6 to 80.6] | 25.0 [0.6 to 80.6] | 40.0 [5.3 to 85.3] | 20.0 [0.5 to 71.6]

4. Secondary Outcome: Percentage of Participants With Polymerase Chain Reaction-adjusted Adequate Clinical and Parasitological Response at Day 42: African <=5 Years PP Population at Day 42 (PP42)
Description: ACPR: negative parasitemia at Day 42, irrespective of AT, in participants not meeting any criteria of ETF: DS or SM at Day 1, 2 or 3 in presence of parasitemia; or Day 2 parasite count > Day 0 irrespective of AT; or parasitemia at Day 3 with AT >=37.5°C; or parasite count on Day 3 >=25% on Day 0, or LCF: DS/ SM in presence of parasitemia between Day 4 and 42; or presence of parasitemia and AT >=37.5°C between Day 4 and 42, or LPF: presence of parasitemia between Day 7 and 42 and AT <37.5°C or having rescue therapy for malaria. PCR-adjusted ACPR was applied to recrudescence (appearance of asexual parasites after clearance of initial infection with a genotype identical to that of parasites present at Baseline), excluding participants with re-infection. Here, in the data table, "overall number of participants analyzed"=participants evaluable for this outcome measure.
Time Frame: Day 42
Population: African <=5 years PP42: participants with parasitologically confirmed Plasmodium falciparum malaria at screening/baseline, received the single administration of OZ439/FQ, without major protocol violations impacting efficacy, evaluable for crude ACPR at Day 42, excluding those who received rescue treatment due to vomiting during drug administration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 43 | 55 | 50 | 57
percentage of participants | 69.8 [53.9 to 82.8] | 81.8 [69.1 to 90.9] | 84.0 [70.9 to 92.8] | 87.7 [76.3 to 94.9]

5. Secondary Outcome: Percentage of Participants With Polymerase Chain Reaction-adjusted Adequate Clinical and Parasitological Response at Day 63: African <=5 Years PP Population at Day 63 (PP63)
Description: ACPR: negative parasitemia at Day 63, irrespective of AT, in participants not meeting any criteria of ETF: DS or SM at Day 1, 2 or 3 in presence of parasitemia; or Day 2 parasite count > Day 0 irrespective of AT; or parasitemia at Day 3 with AT >=37.5°C; or parasite count on Day 3 >=25% on Day 0, or LCF: DS/ SM in presence of parasitemia between Day 4 and 63; or presence of parasitemia and AT >=37.5°C between Day 4 and 63, or LPF: presence of parasitemia between Day 7 and 63 and AT <37.5°C or having rescue therapy for malaria. PCR-adjusted ACPR was applied to recrudescence (appearance of asexual parasites after clearance of initial infection with a genotype identical to that of parasites present at Baseline), excluding participants with re-infection. Here, in the data table, "overall number of participants analyzed"=participants evaluable for this outcome measure.
Time Frame: Day 63
Population: African <=5 years PP63: participants with parasitologically confirmed Plasmodium falciparum malaria at screening/baseline, received the single administration of OZ439/FQ, without major protocol violations impacting efficacy, evaluable for crude ACPR at Day 63, excluding those who received rescue treatment due to vomiting during drug administration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 39 | 43 | 44 | 47
percentage of participants | 64.1 [47.2 to 78.8] | 76.7 [61.4 to 88.2] | 81.8 [67.3 to 91.8] | 87.2 [74.3 to 95.2]

6. Secondary Outcome: Percentage of Participants With Crude Adequate Clinical and Parasitological Response at Day 28: African <=5 Years PP28 Population
Description: ACPR was defined as negative parasitemia at Day 28, irrespective of AT, in participants not meeting any criteria of ETF: DS or SM at Day 1, 2 or 3 in presence of parasitemia; or Day 2 parasite count > Day 0 irrespective of AT; or parasitemia at Day 3 with AT >=37.5°C; or parasite count on Day 3 >=25% on Day 0, or LCF: DS/ SM in presence of parasitemia between Day 4 and 28; or presence of parasitemia and AT >=37.5°C between Day 4 and 28 or, LPF: presence of parasitemia between Day 7 and 28 and AT <37.5°C or having rescue therapy for malaria. PCR-adjusted ACPR applied to recrudescence (appearance of asexual parasites after clearance of initial infection with a genotype identical to that of parasites present at Baseline), excluding participants with re-infection, whereas crude ACPR does not distinguish re-infection (new clone of parasite) or recrudescence.
Time Frame: Day 28
Population: Analysis was performed on African <=5 years PP28 population. Here, "overall number of participants analyzed"=participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 69 | 67 | 63 | 62
percentage of participants | 49.3 [37.0 to 61.6] | 71.6 [59.3 to 82.0] | 76.2 [63.8 to 86.0] | 87.1 [76.1 to 94.3]

7. Secondary Outcome: Percentage of Participants With Crude Adequate Clinical and Parasitological Response at Day 42: African <=5 Years PP42 Population
Description: ACPR was defined as negative parasitemia at Day 42, irrespective of AT, in participants not meeting any criteria of ETF: DS or SM at Day 1, 2 or 3 in presence of parasitemia; or Day 2 parasite count > Day 0 irrespective of AT; or parasitemia at Day 3 with AT >=37.5°C; or parasite count on Day 3 >=25% on Day 0, or LCF: DS/ SM in presence of parasitemia between Day 4 and 42; or presence of parasitemia and AT >=37.5°C between Day 4 and 42 or, LPF: presence of parasitemia between Day 7 and 42 and AT <37.5°C or having rescue therapy for malaria PCR-adjusted ACPR applied to recrudescence (appearance of asexual parasites after clearance of initial infection with a genotype identical to that of parasites present at Baseline), excluding participants with re-infection, whereas crude ACPR did not distinguish re-infection (new clone of parasite) or recrudescence.
Time Frame: Day 42
Population: Analysis was performed on African <=5 years PP42 population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 69 | 65 | 59 | 61
percentage of participants | 39.1 [27.6 to 51.6] | 50.8 [38.1 to 63.4] | 61.0 [47.4 to 73.5] | 68.9 [55.7 to 80.1]

8. Secondary Outcome: Percentage of Participants With Crude Adequate Clinical and Parasitological Response at Day 63: African <=5 Years PP63 Population
Description: Crude ACPR was defined as negative parasitemia at Day 63, irrespective of AT, in participants not meeting any criteria of ETF: DS or SM at Day 1, 2 or 3 in presence of parasitemia; or Day 2 parasite count > Day 0 irrespective of AT; or parasitemia at Day 3 with AT >=37.5°C; or parasite count on Day 3 >=25% on Day 0, or LCF: DS/ SM in presence of parasitemia between Day 4 and 63; or presence of parasitemia and AT >=37.5°C between Day 4 and 63 or, LPF: presence of parasitemia between Day 7 and 63 and AT <37.5°C or having rescue therapy for malaria. PCR-adjusted ACPR applied to recrudescence (appearance of asexual parasites after clearance of initial infection with a genotype identical to that of parasites present at Baseline), excluding participants with re-infection, whereas crude ACPR did not distinguish re-infection (new clone of parasite) or recrudescence.
Time Frame: Day 63
Population: Analysis was performed on African <=5 years PP63 population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 68 | 65 | 59 | 60
percentage of participants | 35.3 [24.1 to 47.8] | 46.2 [33.7 to 59.0] | 57.6 [44.1 to 70.4] | 58.3 [44.9 to 70.9]

9. Secondary Outcome: Time to Re-emergence
Description: Time to re-emergence (in days) was defined as the time to appearance of asexual parasites after clearance of initial infection irrespective of genotype. Participants with no event were censored at the time of study completion, premature study discontinuation, including switch to established anti-malarial treatment or start of any other treatment with anti-malarial activity, whichever was earliest. Re-emergence was confirmed by microscopy (positive blood smear). Kaplan-Maier method was used for estimation. Here, "overall number of participants analyzed"=participants who were included in the analysis of below reported results which consisted of both, who had the event, plus those who were censored.
Time Frame: Up to Day 63
Population: African <=5 years modified Intent-To-Treat (mITT) population: all randomized African participants <=5 years with parasitological confirmed Plasmodium falciparum (P. falciparum) malaria at baseline, who received the single administration of OZ439/FQ and excluding participants who required rescue treatment due to vomiting during drug administration.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 69 | 73 | 70 | 69
days | 36.0 [24.00 to 63.00] | 61.0 [43.00 to NA] — Upper limit of 95% confidence interval (CI) was not estimable due to very low number of participants with the events. | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events. | 64.0 [63.00 to 65.00]

10. Secondary Outcome: Time to Recrudescence
Description: Time to recrudescence (in days) was defined as the time to appearance of asexual parasites after clearance of initial infection with a genotype identical to that of parasites present at Baseline. Recrudescence was confirmed by PCR analysis. Kaplan-Maier method was used for estimation.
Time Frame: Up to Day 63
Population: Analysis was performed on African <=5 years mITT population. Here, "overall number of participants analyzed"=participants who were included in the analysis of below reported results which consisted of both, who had the event, plus those who were censored.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 69 | 73 | 70 | 69
days | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events. | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events. | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events. | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events.

11. Secondary Outcome: Time to Re-infection
Description: Time to re-infection (in days) was defined as the time to appearance of asexual parasites after clearance of initial infection with a genotype that differs from that of parasites present at Baseline. Re-infection was confirmed by PCR analysis. Kaplan-Maier method was used for estimation.
Time Frame: Up to Day 63
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 69 | 73 | 70 | 69
days | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events. | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events. | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events. | 65.0 [NA to NA] — 95% CI was not estimable due to very low number of participants with the events.

12. Secondary Outcome: Parasite Clearance Time (PCT): African <=5 Years PP Population
Description: PCT was defined as the time (in hours) from the start of study drug administration until the time of first negative blood film (no asexual parasites). This first negative film was confirmed by a second negative film which was taken >=6 to <=12 hours of the first film. Kaplan-Meier method was used for the estimation. Here, in the data table "overall number of participants analyzed"=participants who were included in the analysis of below reported results which consisted of both, who had the event, plus those who were censored.
Time Frame: From the start of study drug administration up to the time of the first negative film (up to Day 63)
Population: African<=5years PP population participants with parasitologically confirmed P.falciparum malaria at screening/baseline, received the single administration of OZ439/FQ, without major protocol violation impacting efficacy, evaluable for crude ACPR at pre-defined time point, excluding who had rescue treatment due to vomiting during drug administration
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 69 | 67 | 63 | 62
hours | 36.0 [24.23 to 36.07] | 36.0 [35.93 to 36.10] | 36.1 [36.00 to 48.00] | 36.1 [24.25 to 36.42]

13. Secondary Outcome: Parasite Clearance Time: African >5 Years PP Population
Description: PCT was defined as the time (in hours) from the start of study drug administration until the time of first negative blood film (no asexual parasites). This first negative film was confirmed by a second negative film which was taken >=6 to <=12 hours of the first film. Kaplan-Meier method was used for the estimation. Here, "overall number of participants analyzed"=participants who were included in the analysis of below reported results which consisted of both, who had the event, plus those who were censored.
Time Frame: From the start of study drug administration up to the time of the first negative film (up to Day 63)
Population: African >5years PP population participants with parasitologically confirmed P.falciparum malaria at screening/baseline, received the single administration of OZ439/FQ, without major protocol violation impacting efficacy, evaluable for crude ACPR at pre-defined time point, excluding who had rescue treatment due to vomiting during drug administration
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 11 | 11 | 12 | 10
hours | 24.0 [18.00 to 24.18] | 24.3 [18.07 to 36.00] | 24.3 [12.23 to 36.00] | 27.2 [6.15 to 36.17]

14. Secondary Outcome: Parasite Clearance Time: Asian PP Population
Description: as for outcome 13
Time Frame: From the start of study drug administration up to the time of the first negative film (up to Day 63)
Population: Asian PP population: participants with parasitologically confirmed P.falciparum malaria at screening/baseline, received the single administration of OZ439/FQ, without major protocol violations impacting efficacy, evaluable for crude ACPR at pre-defined time point, excluding who had rescue treatment due to vomiting during drug administration.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 4 | 5 | 5 | 5
hours | 82.0 [79.97 to NA] — Upper limit of 95% CI was not estimable due to very low number of participants with the events. | 75.1 [53.93 to 95.82] | 79.8 [36.00 to NA] — Upper limit of 95% CI was not estimable due to very low number of participants with the events. | 72.2 [60.08 to 79.98]

15. Secondary Outcome: Fever Clearance Time (FCT): African <=5 Years PP Population
Description: FCT was defined as the time (in hours) from start of study drug administration to the first assessment of adjusted body temperature <37.5°C, confirmed by second assessment, taken within >=6 to <=12 hours of the first assessment. Only participants with fever (adjusted body temperature >=37.5°C present at Baseline) and did not receive paracetamol on day of study drug administration until 96 hours after study drug administration were included in FCT analysis. Participants with no event were censored at the time of study completion, premature study discontinuation, including switch to established anti-malarial treatment or start of any other treatment with anti-malarial activity, whichever was earliest. Kaplan-Meier method was used for the estimation.
Time Frame: From the start of study drug administration up to the time of the first temperature measurement <37.5°C (up to Day 63)
Population: Analyzed performed on African <=5 years PP population participants with fever and did not receive paracetamol within 96 hours of study drug administration. Here, "overall number of participants analyzed"=participants who were included in the analysis of below reported results which consisted of both, who had event, plus those who were censored.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 5 | 3 | 4 | 4
hours | 1.0 [1.00 to 24.00] | 1.0 [1.00 to 18.00] | 1.0 [NA to NA] — 95% CI was not estimable as all 4 participants had the same value. | 1.0 [1.00 to 12.00]

16. Secondary Outcome: Fever Clearance Time: African >5 Years PP Population
Description: FCT was defined as the time (in hours) from start of study drug administration to the first assessment of adjusted body temperature <37.5°C, confirmed by second assessment, taken within >=6 to <=12 hours of the first. Only participants with fever (adjusted body temperature >=37.5°C present at Baseline) and did not receive paracetamol on day of study drug administration until 96 hours after study drug administration were included in FCT analysis. Participants with no event were censored at the time of study completion, premature study discontinuation, including switch to established anti-malarial treatment or start of any other treatment with anti-malarial activity, whichever was earliest. Kaplan-Meier method was used for the estimation.
Time Frame: From the start of study drug administration up to the time of the first temperature measurement <37.5°C (up to Day 63)
Population: Analysis was performed on African >5 years PP population participants with fever and did not receive paracetamol within 96 hours of study drug administration. Here, "overall number of participants analyzed"=participants who were included in the analysis of below reported results which consisted of both, who had event, plus those who were censored.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 3 | 1 | 2 | 1
hours | 1.0 [1.00 to 18.00] | 1.0 | 1.5 [1.00 to 2.00] | 2.0

17. Secondary Outcome: Fever Clearance Time: Asian PP Population
Description: FCT was defined as the time (in hours) from start of study drug administration to the first assessment of adjusted body temperature <37.5°C, confirmed by second assessment, taken within >=6 to <=12 hours of the first. Only participants with fever (adjusted body temperature >=37.5°C present at Baseline) and did not receive paracetamol on day of study drug administration until 96 hours after study drug administration were included in FCT analysis. Participants with no event were censored at the time of study completion, premature study discontinuation, including switch to established anti-malarial treatment or start of any other treatment with anti-malarial activity, whichever was earliest. Kaplan-Meier method was used for the estimation. Here, "overall number of participants analyzed"=participants who were included in the analysis of below reported results which consisted of both, who had the event, plus those who were censored.
Time Frame: From the start of study drug administration up to the time of the first temperature measurement <37.5°C (up to Day 63)
Population: Analysis was performed on Asian PP population participants with fever and did not receive paracetamol within 96 hours of study drug administration. Here, '0' in "overall number of participants analyzed"=no participants were evaluable since they had paracetamol within 96 hours of study drug administration.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 1 | 0 | 0 | 1
hours | 18.0 |  |  | 36.0

18. Secondary Outcome: Parasite Reduction Ratio (PRRlog10) at 24 Hours and 48 Hours: African <=5 Years PP Population
Description: The PRR was calculated as the slope of the linear portion of the regression fit of logarithm parasitemia (per milliliter) versus time (in hours). The PRR24 and PRR48 was the drop-in log units over 24 and 48 hours, respectively.
Time Frame: 24 and 48 hours post dose
Population: Analysis was performed on African <=5 years PP population. Here, "overall number of participants analyzed"=participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: ratio
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 63 | 57 | 58 | 53
ratio
  PRR24 (log10) | 2.867 [1.19 to 5.35] | 3.011 [1.10 to 5.63] | 2.397 [1.25 to 4.75] | 2.587 [1.52 to 5.24]
  PRR48 (log10) | 5.734 [2.39 to 10.69] | 6.023 [2.20 to 11.27] | 4.794 [2.50 to 9.50] | 5.174 [3.04 to 10.48]

19. Secondary Outcome: Parasite Reduction Ratio at 24 Hours and 48 Hours: African >5 Years PP Population
Description: as for outcome 18
Time Frame: 24 and 48 hours post dose
Population: Analysis was performed on African >5 years PP population. Here, "overall number of participants analyzed"=participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: ratio
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 7 | 9 | 10 | 8
ratio
  PRR24 (log10) | 2.979 [2.41 to 4.30] | 4.069 [2.16 to 5.00] | 3.288 [2.30 to 4.81] | 3.054 [1.76 to 5.59]
  PRR48 (log10) | 5.957 [4.83 to 8.60] | 8.137 [4.32 to 10.00] | 6.577 [4.61 to 9.63] | 6.108 [3.52 to 11.17]

20. Secondary Outcome: Parasite Reduction Ratio at 24 Hours and 48 Hours: Asian PP Population
Description: as for outcome 18
Time Frame: 24 and 48 hours post dose
Population: Analysis was performed on Asian PP population. Here, "overall number of participants analyzed"=participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: ratio
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 4 | 5 | 4 | 4
ratio
  PRR24 (log10) | 1.167 [1.01 to 1.28] | 1.125 [1.00 to 1.44] | 1.688 [1.07 to 3.12] | 1.353 [1.10 to 1.65]
  PRR48 (log10) | 2.335 [2.03 to 2.56] | 2.250 [1.99 to 2.88] | 3.377 [2.14 to 6.24] | 2.705 [2.21 to 3.31]

21. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Adverse Event of Special Interest (AESI)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had to have a causal relationship with the treatment. SAEs were any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. TEAEs were defined as AEs that developed or worsened or became serious during on-treatment phase that was defined as the time from the start of the first dose of double-blind drug administration up to the Day 63. AE of special interest (AESI) was an AE (serious or non-serious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor was required.
Time Frame: From Baseline up to Day 63
Population: Analyzed on safety population which included all randomized participants who received at least 1 dose or part of a dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 92 | 94 | 96 | 91
Participants
  Any TEAE | 84 | 87 | 85 | 81
  Any treatment-emergent SAE | 0 | 2 | 4 | 2
  Any treatment-emergent AESI | 5 | 8 | 9 | 11
  Any TEAE led to treatment discontinuation | 3 | 2 | 3 | 2
  Any TEAE led to death | 0 | 0 | 0 | 0

22. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax) of Artefenomel
Description: Cmax is the maximum observed plasma concentration of artefenomel.
Time Frame: 2, 4, 6, 12, 24, 48, 72 and 672 hours post dose
Population: Analysis was performed on the PK population for OZ439 which included all participants who received OZ439 and had at least one evaluable blood sample for PK and with adequate documentation of dosing date and sampling date.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 88 | 93 | 93 | 90
nanograms per milliliter | 1072 (95) | 936.7 (91) | 771.8 (92) | 797.8 (119)

23. Secondary Outcome: Pharmacokinetics: Area Under the Curve From Time 0 to Infinity (AUC0-inf) of Artefenomel
Description: Area under the plasma concentration versus time curve from time zero to infinity.
Time Frame: 2, 4, 6, 12, 24, 48, 72 and 672 hours post dose
Population: Analysis was performed on PK population for OZ439.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour per milliliter
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 88 | 93 | 93 | 90
micrograms*hour per milliliter | 14.24 (124) | 12.41 (127) | 9.621 (130) | 9.605 (147)

24. Secondary Outcome: Pharmacokinetics (PK): Apparent Total Clearance of Artefenomel From Plasma After Oral Administration
Description: Clearance is defined as a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: 2, 4, 6, 12, 24, 48, 72 and 672 hours post dose
Population: Focus of PK assessment was to support the analysis of exposure versus efficacy relationship (PK and pharmacodynamic [PD]). Since clearance was considered irrelevant to the objective of the PK and exposure-response analyses, therefore data for this outcome measure were not collected and reported.
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 0 | 0 | 0 | 0

25. Secondary Outcome: Pharmacokinetics: Apparent Volume of Distribution at Steady State After Non-intravenous Administration (Vss/F) of Artefenomel
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: 2, 4, 6, 12, 24, 48, 72 and 672 hours post dose
Population: Focus of PK assessment was to support the analysis of exposure versus efficacy relationship (PK and PD). Since volume of distribution was considered irrelevant to the objective of the PK and exposure-response analyses, therefore data for this outcome measure were not collected and reported.
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 0 | 0 | 0 | 0

26. Secondary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration of Ferroquine (Cmax)
Description: Cmax is the maximum observed plasma concentration of Ferroquine.
Time Frame: 2, 4, 6, 12, 24, 48, 72 and 672 hours post dose
Population: Analysis was performed on the PK population for FQ which included all participants who received FQ and had at least one evaluable blood sample for PK and with adequate documentation of dosing date and sampling date. Here, "overall number of participants analyzed"=participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 88 | 93 | 93 | 90
nanograms per milliliter | 148.1 (52) | 222.8 (66) | 350 (55) | 467.6 (80)

27. Secondary Outcome: Pharmacokinetics: Area Under the Curve From Time 0 to Day 28 (AUC0-day28) of Ferroquine
Description: Area under the plasma concentration versus time curve from time 0 to Day 28 (i.e. 672 hours).
Time Frame: 2, 4, 6, 8, 12, 24, 48, 168, 336 and 672 hours postdose
Population: Analysis was performed on PK population for FQ. Here, "overall number of participants analyzed"=participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour per milliliter
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 88 | 93 | 93 | 90
micrograms*hour per milliliter | 14.92 (40) | 22.56 (48) | 33.84 (48) | 46.4 (52)

28. Secondary Outcome: Pharmacokinetics: Apparent Total Clearance of Ferroquine From Plasma After Oral Administration
Description: Clearance is defined as a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: 2, 4, 6, 12, 24, 48, 72 and 672 hours post dose
Population: Focus of PK assessment was to support the analysis of exposure versus efficacy relationship (PK and PD). Since clearance was considered irrelevant to the objective of the PK and exposure-response analyses, therefore data for this outcome measure were not collected and reported.
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 0 | 0 | 0 | 0

29. Secondary Outcome: Pharmacokinetics: Apparent Volume of Distribution at Steady State After Non-intravenous Administration of Ferroquine
Description: as for outcome 25
Time Frame: 2, 4, 6, 12, 24, 48, 72 and 672 hours post dose
Population: as for outcome 25
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 0 | 0 | 0 | 0

30. Secondary Outcome: Pharmacokinetics: Blood/Plasma Ratio for Ferroquine and Its Active Metabolite SSR97213
Time Frame: 2, 4, 6, 12, 24, 48, 72 and 672 hours post dose
Population: Focus of PK assessment was to support the analysis of exposure versus efficacy relationship (PK and PD). Since blood plasma ratio of active drug and metabolite was considered irrelevant to the objective of the PK and exposure-response analyses, therefore data for this outcome measure were not collected and reported.
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline up to Day 63
Description: Reported AEs were TEAEs, defined as AEs that developed/worsened or became serious during on-treatment phase - defined as the time from the start of the first dose of double-blind drug administration up to Day 63. Analysis was performed on safety population.
Arm/Group | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg)
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/94 | 0/96 | 0/91
Serious Adverse Events (participants affected / at risk) | 0/92 | 2/94 | 4/96 | 2/91
Other Adverse Events (participants affected / at risk) | 77/92 | 79/94 | 77/96 | 74/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) (N=92) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) (N=94) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) (N=96) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg) (N=91)
Malaria (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hepatitis A (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferroquine (up to 400 mg) + Artefenomel (up to 800 mg) (N=92) | Ferroquine (up to 600 mg) + Artefenomel (up to 800 mg) (N=94) | Ferroquine (up to 900 mg) + Artefenomel (up to 800 mg) (N=96) | Ferroquine (up to 1200 mg) + Artefenomel (up to 800 mg) (N=91)
Malaria (Infections and infestations) | 55 (75) | 50 (65) | 40 (49) | 41 (45)
Upper Respiratory Tract Infection (Infections and infestations) | 7 (9) | 6 (8) | 17 (18) | 10 (10)
Bronchitis (Infections and infestations) | 3 (3) | 5 (5) | 4 (4) | 5 (5)
Rhinitis (Infections and infestations) | 4 (4) | 3 (4) | 1 (1) | 7 (8)
Decreased Appetite (Metabolism and nutrition disorders) | 5 (6) | 8 (8) | 5 (5) | 5 (5)
Headache (Nervous system disorders) | 6 (6) | 7 (8) | 7 (8) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 7 (9) | 15 (16) | 15 (17)
Vomiting (Gastrointestinal disorders) | 27 (29) | 27 (28) | 34 (37) | 34 (37)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 11 (12) | 7 (9) | 11 (13)
Abdominal Pain (Gastrointestinal disorders) | 7 (7) | 5 (5) | 5 (5) | 6 (6)
Pyrexia (General disorders) | 7 (9) | 2 (3) | 9 (12) | 10 (10)
Electrocardiogram Qt Prolonged (Investigations) | 6 (6) | 5 (5) | 6 (7) | 8 (8)

LIMITATIONS AND CAVEATS:
The study was terminated early because all treatment arms met the futility criteria for efficacy during the pre-planned interim analysis. On 02-August-2018, recruitment in Asia was stopped due to lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT02497612/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT02497612/SAP_001.pdf